CLINICAL TRIAL: NCT04660019
Title: Combined Scalp and Ear Acupuncture in Patients With Proton Pump Inhibitor- Dependent Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N202004031
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2022-04

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Neurology
Keywords: Acupuncture
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scalp and auricular acupuncture (Experimental): Three scalp acupoints including GV 20, bilateral GB 15, stomach area and four ear acupoints (Shenmen, thalamus, cardia, stomach).
  Interventions: Other: Scalp and auricular acupuncture
- Seed acupressure (Placebo Comparator): Three scalp acupoints including GV 20, bilateral GB 15, stomach area and four ear acupoints (Shenmen, thalamus, cardia, stomach).
  Interventions: Other: Seed acupressure

INTERVENTIONS:
Other: Scalp and auricular acupuncture — Three scalp acupoints including Baihui (GV 20), bilateral Toulinqi (GB 15, stomach area) and four ear acupoints (Shenmen, thalamus, cardia, stomach). The study duration was 2 weeks with four sessions of scalp and auricular acupuncture treatment on day 1, 5, 9 and 14.
  Arms: Scalp and auricular acupuncture
Other: Seed acupressure — Three scalp acupoints including Baihui (GV 20), bilateral Toulinqi (GB 15, stomach area) and four ear acupoints (Shenmen, thalamus, cardia, stomach). The study duration was 2 weeks with four sessions of seed acupressure treatment on day 1, 5, 9 and 14.
  Arms: Seed acupressure

SUMMARY:
According to the statistics of the National Health Insurance Administration Ministry of Health and Welfare, the number of patients about gastroesophageal reflux disease (GERD) has increased from 610,000 to over 760,000 in the past three years (2016-2018). Western medicine mainly uses proton pump inhibitors (PPI) to improve symptoms. For patients who are ineffective in drug treatment, it will be treated by surgical treatment (Laparoscopic Nissen Fundoplication, endoluminal gastroplication).

DETAILED DESCRIPTION:
According to the statistics of the National Health Insurance Administration Ministry of Health and Welfare, the number of patients about gastroesophageal reflux disease (GERD) has increased from 610,000 to over 760,000 in the past three years (2016-2018). Western medicine mainly uses proton pump inhibitors (PPI) to improve symptoms. For patients who are ineffective in drug treatment, it will be treated by surgical treatment (Laparoscopic Nissen Fundoplication, endoluminal gastroplication).

However, it is easy to cause problems such as difficulty swallowing or recurrence postoperatively. In recent years, more and more integrated treatment studies of Chinese and Western medicine have found that acupuncture can improve GERD and can provide patients with another non-surgical treatment. Traditional acupuncture is mainly based on distinguishing diseases (mainly according to Western medicine disease diagnosis, to perform acupoint selection.), dialectics and verification (based on clinical experience, some stimulation areas with outstanding effects on certain symptoms are selected for acupuncture). Acupuncture treatment for GERD primarily utilizes body acupuncture, while scalp and auricular acupuncture for GERD treatment remain scarcely discussed.

This research plan intends to use scalp and auricular acupuncture on recurrent, PPI-dependent GERD and further explore what is the mechanism of acupuncture to improve the symptoms in patients with refractory gastroesophageal reflux. We hypothesized that scalp and auricular acupuncture will reduce scores of reflux disease questionnaire and PPI use compared to placebo treatment with seed acupressure (SAP). If this mechanism can be clarified, it will reduce the patient's overuse of drugs and the cost of surgery in the future, which will be a big boon for Taiwanese health and finances of health insurance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild reflux esophagitis (Los Angeles grades A or B) diagnosed by endoscopy received a 4-month standard-dose PPI therapy and reported the symptoms were improved during the treatment.
* After discontinuing PPI, patients experienced rebound symptoms but quickly found relief upon resuming PPI.

Exclusion Criteria:

* Cannot sign consent form
* Women who are ready to become pregnant or are pregnant.
* Have a history of fainting during acupuncture treatment.
* Those using anticoagulants or antiplatelet agents.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Reflux Diagnostic Questionnaire | One month
  Reflux Diagnostic Questionnaire (RDQ), scores of symptoms of heartburn, dyspepsia, acid regurgitation, and PPI use.
  The participants must have four-time acupuncture/acupressure treatment in two weeks, and each acupuncture/acupressure treatment spends one hour. For the first visit, the participants must write RDQ. After one month, the participants must write RDQ again. The total score is 35 in RDQ; in addition, the minimum score is 7, and the maximum score is 35. The difference in scores will show the effect of treatment. If the first RDQ score is higher than the last RDQ score, it means that the participants' symptom has been improved by acupuncture/acupressure treatment. If the first RDQ score is the same or lower than the last RDQ score, it means the participants' symptom has not been effectively improved by acupuncture/acupressure treatment.
Analysis of cytokines and GABA concentration in blood | Two weeks
  The participants must have four-time acupuncture/acupressure treatment in two weeks, and each acupuncture/acupressure treatment spends one hour. Blood samples were collected before the first time acupuncture/acupressure treatment and after the last acupuncture/acupressure treatment. The differences between cytokines and GABA will help us to understand the possible mechanisms of acupuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shun Wu, PHD, Study Director — Taipei Municipal Wanfang Hospital
Locations (1):
- Wanfang Hospital, Taipei, Wenshan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data is just for combined scalp and auricular acupuncture in patients with proton pump inhibitor- dependent gastroesophageal reflux disease.

REFERENCES:
- [Background] Meining A, Classen M. The role of diet and lifestyle measures in the pathogenesis and treatment of gastroesophageal reflux disease. Am J Gastroenterol. 2000 Oct;95(10):2692-7. doi: 10.1111/j.1572-0241.2000.03175.x. PMID 11051337
- [Background] Scarpellini E, Ang D, Pauwels A, De Santis A, Vanuytsel T, Tack J. Management of refractory typical GERD symptoms. Nat Rev Gastroenterol Hepatol. 2016 May;13(5):281-94. doi: 10.1038/nrgastro.2016.50. Epub 2016 Apr 14. PMID 27075264
- [Background] Gao DX, Bai XH. [Clinical trial of acupuncture treatment of gastroesophageal reflux cough by needling dorsal segment of the Governor Vessel]. Zhen Ci Yan Jiu. 2019 Feb 25;44(2):140-3. doi: 10.13702/j.1000-0607.170761. Chinese. PMID 30945492
- [Background] Sutor AH, Jesdinsky-Buscher C. [Changes in hemostasis during epilespy treatment using dipropyl acetate. Extended study]. Fortschr Med. 1976 Mar 11;94(8):411-4. German. PMID 786839
- [Background] Wolfe JM, Owens DA. Evidence for separable binocular processes differentially affected by artificially induced anisometropia. Am J Optom Physiol Opt. 1979 May;56(5):279-84. doi: 10.1097/00006324-197905000-00001. PMID 495684
- [Background] Mishina Y, Snider TN. Neural crest cell signaling pathways critical to cranial bone development and pathology. Exp Cell Res. 2014 Jul 15;325(2):138-47. doi: 10.1016/j.yexcr.2014.01.019. Epub 2014 Feb 6. PMID 24509233
- [Background] Herisson F, Frodermann V, Courties G, Rohde D, Sun Y, Vandoorne K, Wojtkiewicz GR, Masson GS, Vinegoni C, Kim J, Kim DE, Weissleder R, Swirski FK, Moskowitz MA, Nahrendorf M. Direct vascular channels connect skull bone marrow and the brain surface enabling myeloid cell migration. Nat Neurosci. 2018 Sep;21(9):1209-1217. doi: 10.1038/s41593-018-0213-2. Epub 2018 Aug 27. PMID 30150661
- [Background] Shaw M, Dent J, Beebe T, Junghard O, Wiklund I, Lind T, Johnsson F. The Reflux Disease Questionnaire: a measure for assessment of treatment response in clinical trials. Health Qual Life Outcomes. 2008 Apr 30;6:31. doi: 10.1186/1477-7525-6-31. PMID 18447946
- [Background] Zanella AK, Gutierres JM, Stigger F. Effects of Scalp Acupuncture on Functional Deficits Induced by Early Sensorimotor Restriction. J Acupunct Meridian Stud. 2019 Jun;12(3):77-83. doi: 10.1016/j.jams.2019.03.002. Epub 2019 Apr 24. PMID 31028972
- [Background] Kattalai Kailasam V, Anand P, Melyan Z. Establishing an animal model for National Acupuncture Detoxification Association (NADA) auricular acupuncture protocol. Neurosci Lett. 2016 Jun 15;624:29-33. doi: 10.1016/j.neulet.2016.05.001. Epub 2016 May 4. PMID 27155456